CLINICAL TRIAL: NCT04033458
Title: A Randomized, Open-Label, 5-way Crossover Study in Healthy Male Participants to Evaluate the Bioavailability, Food Effect, Safety and Tolerability of Two Oral Solid Dosage Formulations Relative to an Oral Solution Formulation of JNJ-64140284.
Brief Title: A Study of JNJ-64140284 Solid Dose Formulations in Healthy Male Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: stopped because of a business decision
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR108648; 2019-001975-35 (EudraCT Number); 64140284EDI1004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Treatment Sequence ABECD (Experimental): Participants will receive single oral dose of JNJ-64140284 Regimen 1 in fasted condition (Treatment A) followed by JNJ-64140284 Regimen 2 in fasted condition (Treatment B), then JNJ-64140284 Regimen 5 in fed condition (Treatment E) followed by JNJ-64140284 Regimen 3 in fed condition (Treatment C) and, then JNJ-64140284 Regimen 4 in fed condition (Treatment D) in Treatment Periods 1 to 5 respectively. All treatment periods will be separated by a wash out period of at least 5 days and maximally 12 days.
  Interventions: Drug: JNJ-64140284
- Treatment Sequence BCADE (Experimental): Participants will receive single oral dose of JNJ-64140284 Regimen 2 in fasted condition (Treatment B) followed by JNJ-64140284 Regimen 3 in fed condition (Treatment C) then JNJ-64140284 Regimen 1 in fasted condition (Treatment A) followed by JNJ-64140284 Regimen 4 in fed condition (Treatment D) and, then JNJ-64140284 Regimen 5 in fed condition (Treatment E) in Treatment Periods 1 to 5 respectively. All treatment periods will be separated by a wash out period of at least 5 days and maximally 12 days.
  Interventions: Drug: JNJ-64140284
- Treatment Sequence CDBEA (Experimental): Participants will receive single oral dose of JNJ-64140284 Regimen 3 in fed condition (Treatment C) followed by JNJ-64140284 Regimen 4 in fed condition (Treatment D) then, JNJ-64140284 Regimen 2 in fasted condition (Treatment B) followed by JNJ-64140284 Regimen 5 in fed condition (Treatment E) and then, JNJ-64140284 Regimen 1 in fasted condition (Treatment A) in Treatment Periods 1 to 5 respectively. All treatment periods will be separated by a wash out period of at least 5 days and maximally 12 days.
  Interventions: Drug: JNJ-64140284
- Treatment Sequence DECAB (Experimental): Participants will receive single oral dose of JNJ-64140284 Regimen 4 in fed condition (Treatment D) followed by JNJ-64140284 Regimen 5 in fed condition (Treatment E) then JNJ-64140284 Regimen 3 in fed condition (Treatment C) followed by JNJ-64140284 Regiment 1 in fasted condition (Treatment A) and then JNJ-64140284 Regimen 2 in fasted condition (Treatment B) in Treatment Periods 1 to 5 respectively. All treatment periods will be separated by a wash out period of at least 5 days and maximally 12 days.
  Interventions: Drug: JNJ-64140284
- Treatment Sequence EADBC (Experimental): Participants will receive single oral dose of JNJ-64140284 Regimen 5 in fed condition (Treatment E) followed by JNJ-64140284 Regimen 1 in fasted condition (Treatment A) then JNJ-64140284 Regimen 4 in fed condition (Treatment D) then JNJ-64140284 Regimen 2 in fasted condition (Treatment B) and then, JNJ-64140284 Regimen 3 in fed condition (Treatment C) in Treatment Periods 1 to 5 respectively. All treatment periods will be separated by a wash out period of at least 5 days and maximally 12 days.
  Interventions: Drug: JNJ-64140284
- Treatment Sequence DCEBA (Experimental): Participants will receive single oral dose of JNJ-64140284 Regimen 4 in fed condition (Treatment D) followed by JNJ-64140284 Regimen 3 in fed condition (Treatment C) then JNJ-64140284 Regimen 5 in fed condition (Treatment E) followed by JNJ-64140284 Regimen 2 in fasted condition (Treatment B) and then JNJ-64140284 Regimen 1 in fasted condition (Treatment A) in Treatment Periods 1 to 5 respectively. All treatment periods will be separated by a wash out period of at least 5 days and maximally 12 days.
  Interventions: Drug: JNJ-64140284
- Treatment Sequence EDACB (Experimental): Participants will receive single oral dose of JNJ-64140284 Regimen 5 in fed condition (Treatment E) followed by JNJ-64140284 Regimen 4 in fed condition (Treatment D) then JNJ-64140284 Regimen 1 in fasted condition (Treatment A) followed by JNJ-64140284 Regimen 3 in fed condition (Treatment C) and then JNJ-64140284 Regimen 2 in fasted condition (Treatment B) in Treatment Periods 1 to 5 respectively. All treatment periods will be separated by a wash out period of at least 5 days and maximally 12 days.
  Interventions: Drug: JNJ-64140284
- Treatment Sequence AEBDC (Experimental): Participants will receive single oral dose of JNJ-64140284 Regimen 1 in fasted condition (Treatment A) followed by JNJ-64140284 Regimen 5 in fed condition (Treatment E) then JNJ-64140284 Regimen 2 in fasted condition (Treatment B) followed by JNJ-64140284 Regimen 4 in fed condition (Treatment D) and then JNJ-64140284 Regimen 3 in fed condition (Treatment C) in Treatment Periods 1 to 5 respectively. All treatment periods will be separated by a wash out period of at least 5 days and maximally 12 days.
  Interventions: Drug: JNJ-64140284
- Treatment Sequence BACED (Experimental): Participants will receive single oral dose of JNJ-64140284 Regimen 2 in fasted condition (Treatment B) followed by JNJ-64140284 Regimen 1 in fasted condition (Treatment A) then JNJ-64140284 Regimen 3 in fed condition (Treatment C) followed by JNJ-64140284 Regimen 5 in fed condition (Treatment E) and then JNJ-64140284 Regimen 4 in fed condition (Treatment D) in Treatment Periods 1 to 5 respectively. All treatment periods will be separated by a wash out period of at least 5 days and maximally 12 days.
  Interventions: Drug: JNJ-64140284
- Treatment Sequence CBDAE (Experimental): Participants will receive single oral dose of JNJ-64140284 Regimen 3 in fed condition (Treatment C) followed by JNJ-64140284 Regimen 2 in fasted condition (Treatment B) then JNJ-64140284 Regimen 4 in fed condition (Treatment D) followed by JNJ-64140284 Regimen 1 in fasted condition (Treatment A) and then JNJ-64140284 Regimen 5 in fed condition (Treatment E) in Treatment Periods 1 to 5 respectively. All treatment periods will be separated by a wash out period of at least 5 days and maximally 12 days.
  Interventions: Drug: JNJ-64140284

INTERVENTIONS:
Drug: JNJ-64140284 — Participants will receive JNJ-64140284 orally.
  Other Names: AMPARγ8

SUMMARY:
The purpose of this study is to compare the pharmacokinetic profile of a single dose of two solid dosage formulations relative to a reference formulation (solution in polyethylene glycol-400 [PEG-400]) of JNJ-64140284 in healthy male participants under fasting condition and to assess the effect of food on the bioavailability of two solid dosage formulations of JNJ-64140284.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 18.0 and 29.9 kilograms per square meter (kg/m^2) inclusive
* Participants must be healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, retesting of an abnormal lab value(s) that may lead to exclusion will be allowed once during the screening phase. The participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study according to the investigator. This determination must be recorded in the participant's source documents and initialed by the investigator
* Participant must be healthy on the basis of physical examination, medical history, vital signs, and 12-lead Electrocardiogram (ECG) (means of triplicate ECG, inclusive QTcF less than or equal to [<=] 450 milliseconds [msec]) performed at screening and admission to the clinical unit. Minor abnormalities in ECG, which are not considered to be of clinical significance by the investigator, are acceptable. The presence of left bundle branch block (LBBB), atrioventricular (AV) block (second degree or higher), or a permanent pacemaker or implantable cardioverter defibrillator [ICD] will lead to exclusion
* Non-smokers (not smoked cigarettes or equivalent or not used nicotine-based products for 3 months prior to screening)
* Men who are sexually active with a woman of childbearing potential and have not had a vasectomy must agree to use a barrier method of birth control for example, either condom or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository for the duration of the study plus 3 months after receiving the last dose of study drug, and all men must not donate sperm during the study and for 3 months after receiving the last dose of study drug. In addition, their female partners should also use an additional method of birth control (which may include a hormonal method, an intrauterine device [IUD] or an intrauterine system [IUS]) for at least the same duration. Men with a partner who is pregnant, you must use a condom to avoid exposure to the unborn child

Exclusion Criteria:

* History of or current significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematological disease, lipid abnormalities, bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, Parkinson's disease, infection, or any other illness that the Investigator considers should exclude the participant
* Serology positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies or human immunodeficiency virus (HIV) antibodies
* Participant has a history of at least mild drug or alcohol use disorder according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-V) criteria within 6 months before Screening or positive test result(s) for alcohol and/or drugs of abuse (opiates (including methadone), cocaine, amphetamines, methamphetamines, cannabinoids, barbiturates, ecstasy and benzodiazepines) at screening or admission
* Drinks, on average, more than 5 cups of tea or coffee or 8 cans of cola per day
* Clinically significant acute illness within 7 days prior to study drug administration

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of JNJ-64140284 | Predose, 0.25, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36 and 48 hours postdose
  Cmax is defined as the peak plasma concentration of JNJ-64140284.
Area Under The Plasma Concentration-time Curve From 0 to t Hours Postdosing (AUC[0-t]) of JNJ-64140284 | Predose, 0.25, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36 and 48 hours postdose
  AUC(0-t) is defined as the area under the plasma concentration-time curve from 0 to t hours postdosing of JNJ-64140284 (time t is the time of the last quantifiable concentration [Clast]).
Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC[0-inf]) of JNJ-64140284 | Predose, 0.25, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36 and 48 hours postdose
  AUC(0-inf) is defined as the area under plasma concentration-time from time 0 to infinity extrapolated to infinity of JNJ-64140284.
Relative Bioavailability (F[rel]) of JNJ-64140284 | Predose, 0.25, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36 and 48 hours postdose
  F(rel) is defined as the relative bio-availability of JNJ-64140284 calculated as individual Cmax and AUC treatment ratio's (for the comparison of the capsule [solid 5 micro-meter (mcm) or solid 31 mcm] to the solution and for the comparison of fed versus fasted for the capsule [both for solid 5 mcm and solid 31 mcm]).

SECONDARY OUTCOMES:
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Up to 13 weeks
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency